CLINICAL TRIAL: NCT06485765
Title: The Effect of the DASH (Dietary Approaches to Stop Hypertension) Diet on Quality of Life and Cardiac Parameters in Patients Acute Coronary Syndrome With Hypertension
Brief Title: DASH Diet, Quality of Life and Cardiac Parameters of Patients With Acute Coronary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Hacı Ömer YILMAZ, Assistant Professor (PhD), Bandırma Onyedi Eylül University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: hcmrylmz-2024
Record Dates: First submitted 2024-06-17; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Acute Coronary Syndrome; Hypertension
Keywords: acute coronary syndrome; hypertension; DASH diet; quality of life; cardiac parameters
MeSH Terms: conditions — Acute Coronary Syndrome; Hypertension

STUDY DESIGN:
Intervention Model Description: This clinical trial is a single-group, pre-post design. In this model, quality of life and cardiac parameters were assessed before and after individualised DASH diet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): The daily energy requirement of the individuals included in the study was obtained by multiplying the physical activity level (PAL) calculated as a result of 24-hour physical activity recording and the Harris-Benedict formula used to calculate the basal metabolic rate.
  Harris-Benedict Formula Male 66.5 + 13.75 x Weight (kg) + 5.003 x Height (cm) - 6.775 x Age (years) Female 655.1 + 9.563 x Weight (kg) + 1.85 x Height (cm) - 4.676 x Age (years)
  After the daily energy requirement was calculated, a DASH eating plan specific to the individuals was created and they were asked to maintain it for 12 weeks. In addition, the personal contact information of the researcher was shared with the individuals and they were in constant communication about all questions related to the nutrition plan.
  Interventions: Other: Diet planning

INTERVENTIONS:
Other: Diet planning — Healthy eating planning

SUMMARY:
The clinical trail study aimed to determine effect of DASH eating plan on cardiac parameters and quality of life in hypertensive individuals diagnosed with acute coronary syndrome.

The main questions it aims to answer are:

1. DASH diet improve quality of life?
2. DASH diet improve cardiac parameters?

The researchers assessed the results of 12 weeks of the DASH diet.

Patients will apply the DASH diet prepared individually by the researchers for 12 weeks.

DETAILED DESCRIPTION:
The study period was 12 weeks. Patients' food consumption (3 day), anthropometric measurements, blood pressure measurements, physical activity levels, biochemical and cardiac parameters, adherence to DASH eating plan and the MacNew Heart Health-Related Quality of Life Scale were recorded at the beginning of the study and at the end of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with acute coronary syndrome within the last month
* with a measured blood pressure above 140/90 mmHg or using antihypertensive drugs
* not obese (body mass index < 30)
* not diagnosed with a disease requiring a different medical nutrition therapy (chronic renal failure, diabetes, cancer, etc.)
* volunteered to participate in the study

Exclusion Criteria:

* Acute coronary syndrome diagnosed more than 1 month ago
* obese (body mass index > 30 )
* without hypertension
* receiving different medical nutrition therapy

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Quality of Life (MacNew Heart Disease Health-Related Quality of Life Scale) | 12 week
  The quality of life of the patients at the beginning of the study and at the end of the 12th week was assessed with the MacNew Heart Disease Health-Related Quality of Life Scale. The scale is a different form of the Post-MI Quality of Life Scale, which was developed to determine especially depression and anxiety in patients with acute MI (Myocardial Infarction) and which can be evaluated by patients responding to the scale. The scale can be used in different cardiac patients such as MI, angina pectoris and heart failure patients and there is a high correlation between it and other tools that assess quality of life. MacNew Heart Disease Health-Related Quality of Life Scale consists of three sub-dimensions (emotional, physical and social) and 27 items in 7-point Likert type. The answer to each item is between 1-7. A low score indicates poor quality of life, while a high score indicates better quality of life.
Ejection Fraction (%) | 12 weeks
  A measurement of the percentage of blood leaving the heart each time it squeezes (using echocardiographic imaging)

CONTACTS AND LOCATIONS:
Locations (1):
- Bandırma Onyedi Eylul University, Balıkesir, Bandırma, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared after the data is obtained and analysed
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12 months